CLINICAL TRIAL: NCT03963076
Title: Evaluation of the Efficiency of Nasal Spray Hypertonic Puressentiel on Symptoms of Patients With Allergic Rhinitis
Brief Title: Efficacy of Nasal Spray Hypertonic Puressentiel on Symptoms of Allergic Rhinitis
Acronym: ENAPAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Puressentiel (Industry)
Collaborators: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Puressentiel
Record Dates: First submitted 2019-05-18; First posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Oils, Volatile

STUDY DESIGN:
Intervention Model Description: prospective multicentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- allergic rhinitis (Experimental): administration of a nasal hypertonic spray twice a day for one month
  Interventions: Other: nasal hypertonic spray: combination of hypertonic sea water and organic rosemary floral water with essential oils (ravintsara, geranium, eucalyptus radiata, niaouli)

INTERVENTIONS:
Other: nasal hypertonic spray: combination of hypertonic sea water and organic rosemary floral water with essential oils (ravintsara, geranium, eucalyptus radiata, niaouli) — One spray of nasal hypertonic spray morning and evening every day during 30 days

SUMMARY:
Prospective multicentric study.

60 subjects with allergic rhinitis will be enrolled to test the efficacy of nasal hypertonic spray Puressentiel on symptoms of allergic rhinitis and nasal peak flow.

Subjects with allergic rhinitis and nasal obstruction will use during 30 days the nasal spray (2 nebulisations /day in each nostril) during 30 days.

Rhinitis symptoms questionnaire and nasal inspiratory peak flow will be evaluated before and after 30 days of exposure.

DETAILED DESCRIPTION:
Objective: evaluate the efficiency of a nasal hypertonic spray Puressentiel in subjects with allergic rhinitis and nasal obstruction.

Inclusion criteria: subjects with allergic obstructive rhinitis without treatment or remaining symptomatic despite treatment.

Duration of exposure: 2 nasal sprays per day (morning and evening) during 30 months.

Primary criteria of efficacy: Rhinitis questionnaire.

Secondary criteria: Inspiratory nasal peak flow

ELIGIBILITY:
Inclusion Criteria:

* allergic rhinitis with nasal obstruction

Exclusion Criteria:

* pregnant patients
* patients with severe asthma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Rhinitis auto questionnaire symptoms | Measurement at Day 0
  5 questions quoted from 1 (worse) to 5 (best).
Rhinitis auto questionnaire symptoms | Measurement at Day 30
  5 questions quoted from 1 (worse) to 5 (best).

SECONDARY OUTCOMES:
Nasal inspiratory peak flow | Measurement at Day 0 and Day 30
  Inspiratory nasal peak flow
Nasal inspiratory peak flow | Measurement at Day 30
  Inspiratory nasal peak flow

CONTACTS AND LOCATIONS:
Locations (1):
- Caroline Bonnard, Paris, France

IPD SHARING:
Plan to Share IPD: No